CLINICAL TRIAL: NCT02260999
Title: Experimental Study of Detection an Intentional Performance Degradation in Grip Strength
Status: Completed | Type: Observational
Sponsor: Christoph Maier, Prof. Dr. (Other)
Responsible Party: Sponsor-Investigator, Christoph Maier, Prof. Dr., Prof. Dr.med. C. Maier, Ruhr University of Bochum
Organization: Ruhr University of Bochum (Other)
Other Study IDs: BHL-2113
Record Dates: First submitted 2014-10-06; First posted 2014-10-09 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- healthy: > 18 years old sufficient language knowledge
- chronic pain patients
- patients with injury at the upper etxremity

SUMMARY:
In this study, the detection of the feigning weakness in grip strength is measured using different grip strength testing instruments. Patients with injury of the upper limb are compared to patients with injury of the lower limb as well as healthy controls.

ELIGIBILITY:
Inclusion Criteria:

- >18 years, signed consent form, stable pain mediaction for 48 hours

Exclusion Criteria:

- <18, unsigned consent form, dose change of the pain medication during the last 48 hours...

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: chronic pain patients patients with injury at the upper extremity healthy subjects
Sampling Method: Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2012-05; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
grip strength | 1 hour
  mean and maximum grip strength measured by rapid exchange grip and isometric grip strength testing
range of motion | 1 hour
  measured by the handtutor